CLINICAL TRIAL: NCT01877382
Title: A Phase 1 Multiple Ascending Dose Study of Milademetan in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: A Multiple Ascending Dose Study of Milademetan in Subjects With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3032-A-U101
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — milademetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1, Milademetan Alone (Experimental): Participants receive milademetan alone with different dose schedules.
  Interventions: Drug: Milademetan
- Part 2, Milademetan Alone (Experimental): Participants with advanced melanoma and diffuse large B cell lymphoma (DLBCL) receive milademetan alone with different dose schedules.
  Interventions: Drug: Milademetan

INTERVENTIONS:
Drug: Milademetan — DS-3032b will be administered as an oral capsule. It will be supplied in 5, 20, 80, and/or 200 mg capsules individually packaged in desiccant-embedded aluminum blisters.
  Arms: Part 1, Milademetan Alone
Drug: Milademetan — Milademetan will be administered as a single oral capsule or as a combination of multiple oral capsules containing 5, 20, 80, and/or 200 mg. An alternate combination of 30 and/or 100 mg capsules of milademetan may be utilized.
  Arms: Part 2, Milademetan Alone

SUMMARY:
This will be a Phase 1, open-label study of milademetan to assess its safety and tolerability, identify a maximum tolerated dose (MTD)/tentative recommended phase 2 dose (RP2D), and assess its pharmacokinetic (PK)/ pharmacodynamic (PDy) properties in participants with advanced solid tumors or lymphomas.

Approximately 5 US sites are planned for Part 1 (Dose Escalation) and Part 2 (Dose Expansion). The same sites are planned to participate for both parts.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Cohorts (Part 1)

* Has a histologically or cytologically documented advanced solid tumor or lymphoma that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available.

  * Participants with melanoma who are ineligible to receive or have declined ipilimumab treatment or who are refractory or intolerant to ipilimumab may enroll.
  * Participants with certain tumor types such as those with high prevalence of MDM2 amplification or overexpression (eg, well-differentiated [WD]/dedifferentiated [DD] liposarcoma) may be preferentially enrolled in Part 1.

Dose Expansion Cohort (Part 2)

* Has a histologically or cytologically documented advanced melanoma or diffuse large B cell lymphoma (DLBCL), with measurable disease that is refractory to standard treatment or for which no standard treatment is available.

  * Participants with melanoma who are ineligible to receive or have declined ipilimumab treatment or who are refractory or intolerant to ipilimumab may enroll.
  * Participants with DLBCL who have failed, been deemed ineligible for, or refused autologous stem cell transplantation may enroll.
* Man or woman ≥ 18 years old.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Has adequate bone marrow function, defined as:

  * Platelet count ≥ 100 x 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1.5 x 10^9/L.
* Has adequate renal function, defined as creatinine clearance ≥ 60 mL/min, as calculated using the modified Cockcroft Gault equation, ([{140 - age in years} × {actual weight in kg}] divided by [{72 × serum creatinine in mg/dL} multiply by 0.85 if female]), OR creatinine ≤ 1.5 x ULN.
* Has adequate hepatic function, defined as:

  * AST/ALT levels ≤ 3 x ULN (if liver metastases are present, ≤ 5 x ULN)
  * Bilirubin ≤ 1.5 x ULN.
* Has adequate blood clotting function, defined as International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
* Participant should be able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or comorbidity that would interfere with therapy.
* Participant (male and female) of childbearing/reproductive potential must agree to use double-barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug.
* Participant must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IRB [Institutional Review Board]-approved Informed consent Form [ICF] (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study specific procedures or tests.
* Is willing to provide and there is confirmed availability of pre-existing diagnostic or resected tumor samples, such as paraffin-embedded sections. Providing fresh tumor biopsy is optional for participants in Dose Escalation cohorts.
* Is willing to undergo tumor genotyping for TP53 mutation, insertion, or deletion at screening. Confirmation of TP53 nonmutant status is encouraged, but not required prior to milademetan dosing.
* Is willing to provide additional archived samples for comprehensive genomic and/or proteomic analyses if the participant has a partial response/complete response to milademetan treatment.
* Is willing to undergo pre-treatment tumor biopsies (Part 2 only)

Exclusion Criteria:

* Has a tumor that contains an inactivating mutation, insertion, or deletion in the TP53 gene determined previously or at screening.
* Has a history of primary central nervous system malignancy.
* Has gastrointestinal conditions that could affect the absorption of milademetan in the opinion of the Investigator.
* Has an uncontrolled infection requiring intravenous antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or active hepatitis B or C infection.
* Has received an allogeneic bone marrow or allogeneic stem cell transplant.
* Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor.
* Has clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (2 weeks for stereotactic radiotherapy).
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE v4, grade ≤ 1 or baseline. Participants with chronic grade 2 toxicities may be eligible per the discretion of the Investigator and Sponsor (eg, grade 2 chemotherapy-induced neuropathy).
* Had an autologous transplant within 3 months of starting study drug treatment.
* Is receiving concomitant treatment with a strong inducer of CYP3A.
* Had systemic treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy within 3 weeks before study drug treatment; or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment; or treatment with small-molecule targeted agents within 2 weeks before study drug treatment. Previous and concurrent use of hormone replacement therapy, the use of gonadotropin releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted if such therapy has not been changed within 8 weeks before study drug treatment.
* Had therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment.
* Participated in a therapeutic clinical study within 3 weeks before study drug treatment, or current participation in other therapeutic investigational procedures.
* Prolongation of corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is > 450 milliseconds (ms) for males and > 470 ms for females based on triplicate ECG.
* Pregnant or breastfeeding.
* Substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the participant's participation in the clinical study or evaluation of the clinical study results.
* Prior treatment with an MDM2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (5):
- United States (5):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University College of Physicians and Surgeons, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Gounder MM, Bauer TM, Schwartz GK, Weise AM, LoRusso P, Kumar P, Tao B, Hong Y, Patel P, Lu Y, Lesegretain A, Tirunagaru VG, Xu F, Doebele RC, Hong DS. A First-in-Human Phase I Study of Milademetan, an MDM2 Inhibitor, in Patients With Advanced Liposarcoma, Solid Tumors, or Lymphomas. J Clin Oncol. 2023 Mar 20;41(9):1714-1724. doi: 10.1200/JCO.22.01285. Epub 2023 Jan 20. PMID 36669146
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36669146/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 participants who met all inclusion criteria and no exclusion criteria were enrolled and received treatment.
Pre-assignment Details: Dose escalation of milademetan to determine the maximum tolerated dose started with an initial accelerated titration design and then switched to a Bayesian logistic regression model with escalation with overdose control.
Groups:
- Cohort 1: 15 mg/Day Milademetan: Participants who received 15 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 2: 30 mg/Day Milademetan: Participants who received 30 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 3: 60 mg/Day Milademetan: Participants who received 60 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 4: 120 mg/Day Milademetan; Expansion Cohort: 120 mg/Day Milademetan: Participants who received 120 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 5: 240 mg/Day Milademetan: Participants who received 240 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 6: 160 mg/Day Milademetan: Participants who received 160 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 7b: 90 mg/Day Milademetan: Participants who received 90 mg/day milademetan daily (QD) x 28/28 days.
- Cohort 8c: 90 mg/Day Milademetan: Participants who received 90 mg/day milademetan daily (QD) x 21/28 days.
- Cohort 9d: 120 mg/Day Milademetan: Participants who received 120 mg/day milademetan daily (QD) x 7/28 days.
- Cohort 10e: 120 mg/Day Milademetan: Participants who received 120 mg/day milademetan daily (QD) x 3/14 days x 2 in a 28-day cycle.
- Cohort 11e: 200 mg/Day Milademetan: Participants who received 200 mg/day milademetan daily (QD) x 3/14 days x 2 in a 28-day cycle.
- Cohort 12d: 200 mg/Day Milademetan: Participants who received 200 mg/day milademetan daily (QD) x 7/28 days.
- Cohort 13e: 260 mg/Day Milademetan: Participants who received 260 mg/day milademetan daily (QD) x 3/14 days x 2 in a 28-day cycle.
- Cohort 14e: 340 mg/Day Milademetan: Participants who received 340 mg/day milademetan daily (QD) x 3/14 days x 2 in a 28-day cycle.
Period: Dose Escalation
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan | Expansion Cohort: 120 mg/Day Milademetan
Started | 3 | 1 | 1 | 13 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 1 | 13 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3 | 0
Not completed — Progressive disease | 2 | 0 | 1 | 6 | 1 | 0 | 3 | 10 | 4 | 2 | 3 | 3 | 13 | 1 | 0
Not completed — TP53 gene nonsynonymous mutation, insertion, or deletion detected | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical progression | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Period: Dose Expansion
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan | Expansion Cohort: 120 mg/Day Milademetan
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — TP53 gene nonsynonymous mutation, insertion, or deletion detected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan | Expansion Cohort: 120 mg/Day Milademetan | Total
Number analyzed (Participants) | 3 | 1 | 1 | 13 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3 | 20 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 0 | 11 | 2 | 2 | 5 | 8 | 5 | 2 | 2 | 3 | 15 | 3 | 10 | 71
  >=65 years | 0 | 1 | 1 | 2 | 0 | 3 | 4 | 7 | 1 | 1 | 1 | 0 | 5 | 0 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (0) | 69.0 | 67.0 | 59.8 (8.6) | 55.0 (12.7) | 64.0 (10.9) | 59.0 (12.0) | 63.4 (12.0) | 55.8 (11.1) | 53.3 (15.8) | 56.0 (28.2) | 46.0 (5.6) | 58.9 (11.4) | 57.3 (2.9) | 61.3 (12.4) | 59.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 7 | 2 | 4 | 4 | 9 | 3 | 1 | 1 | 2 | 8 | 2 | 8 | 53
  Male | 1 | 1 | 1 | 6 | 0 | 1 | 5 | 6 | 3 | 2 | 2 | 1 | 12 | 1 | 12 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 6
  White | 2 | 1 | 1 | 12 | 0 | 4 | 9 | 15 | 4 | 3 | 2 | 2 | 16 | 2 | 17 | 90
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 1 | 13 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3 | 20 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (≥10% Overall) in Participants Receiving Milademetan
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that emerged during the treatment period (from first dose date until 30 days after the last dosing date), having been absent at pretreatment; or reemerged during treatment, having been present at baseline, but stopped prior to treatment; or worsened in severity after starting treatment relative to the pretreatment state, when the AE was continuous.
Time Frame: Screening until end of treatment visit, up to approximately 7 years 2 months
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4: 120 mg/Day Milademetan + Expansion Cohort: Participants who received 120 mg/day milademetan daily (QD) x 21/28 days.
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 33 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3
Participants
  Any TEAE | 3 | 1 | 1 | 33 | 2 | 5 | 9 | 15 | 6 | 3 | 3 | 3 | 20 | 3
  Nausea | 1 | 0 | 0 | 22 | 2 | 5 | 7 | 13 | 4 | 1 | 2 | 3 | 16 | 2
  Diarrhea | 0 | 0 | 0 | 16 | 1 | 3 | 4 | 7 | 0 | 1 | 1 | 1 | 9 | 2
  Vomiting | 1 | 0 | 0 | 10 | 2 | 3 | 2 | 4 | 2 | 1 | 1 | 1 | 11 | 2
  Constipation | 1 | 0 | 0 | 7 | 1 | 0 | 4 | 5 | 2 | 1 | 1 | 0 | 5 | 0
  Abdominal pain | 1 | 0 | 0 | 5 | 0 | 2 | 1 | 4 | 0 | 1 | 0 | 0 | 3 | 1
  Thrombocytopenia | 0 | 0 | 0 | 25 | 1 | 4 | 5 | 13 | 2 | 1 | 1 | 2 | 11 | 2
  Anemia | 1 | 0 | 1 | 16 | 1 | 3 | 4 | 9 | 2 | 0 | 2 | 2 | 5 | 0
  Leukopenia | 0 | 0 | 0 | 9 | 1 | 5 | 5 | 9 | 1 | 1 | 1 | 0 | 7 | 0
  Neutropenia | 0 | 0 | 0 | 9 | 1 | 4 | 4 | 6 | 1 | 0 | 0 | 0 | 4 | 0
  Lymphopenia | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 2 | 0 | 4 | 0
  Fatigue | 0 | 0 | 0 | 18 | 2 | 4 | 4 | 10 | 4 | 2 | 1 | 2 | 10 | 2
  Edema peripheral | 2 | 0 | 0 | 4 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 1 | 3 | 0
  Pyrexia | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 3 | 0
  Decreased appetite | 1 | 0 | 0 | 10 | 2 | 5 | 5 | 7 | 1 | 1 | 0 | 0 | 8 | 2
  Dyspnea | 1 | 0 | 0 | 5 | 1 | 1 | 2 | 5 | 3 | 0 | 0 | 0 | 4 | 0
  Cough | 1 | 0 | 0 | 4 | 0 | 2 | 3 | 6 | 1 | 0 | 0 | 1 | 3 | 0
  Dysgeusia | 1 | 0 | 0 | 7 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 4 | 0
  Headache | 0 | 0 | 0 | 5 | 1 | 1 | 2 | 4 | 2 | 1 | 0 | 0 | 2 | 1
  Aspartate aminotransferase increased | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities In Participants Receiving Milademetan by Preferred Term and Worst Grade by NCI CTCAE
Description: A dose-limiting toxicity (DLT) was defined as any treatment-emergent AE (TEAE) not attributable to the participant's disease or a disease-related processes that occurred during the observation period (Cycle 1) in each dose-level cohort and was Grade 3 or higher according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0, with a few exceptions.
Time Frame: Cycle 1, Day 1 to Day 28 (each cycle, 28 days)
Population: Dose-limiting toxicities were assessed in the DLT Evaluable Set in cohorts with available patient data. DLTs were not evaluated in the Expansion Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 2 | 1 | 1 | 13 | 1 | 5 | 8 | 15 | 6 | 3 | 3 | 3 | 18 | 3
Participants
  Any TEAE classified as DLT | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Grade 4 DLT | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 DLT | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 DLT | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Thrombocytopenia | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 4 Thrombocytopenia | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Thrombocytopenia | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Leukopenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Neutropenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Nausea | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Malaise | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Malaise | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Decreased appetite | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Decreased appetite | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Melanoma and Diffuse Large B Cell Lymphoma Who Achieved Objective Response
Description: Tumor response was assessed using RECIST Version 1.1 (in solid tumor participants with measurable disease) or treatment response using the revised International Working Group criteria 7 (in participants with lymphoma). For RECIST, complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Objective response rate (ORR) was the sum of CR and PR rates.
Time Frame: Screening up to Cycle 3 and beyond, Day 1 (each cycle, 28 days)
Population: Objective response was assessed in the Dose Expansion cohort of the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: 120 mg/Day Milademetan
Number analyzed (Participants) | 20
Participants
  Complete response | 0
  Partial response | 1
  Stable disease | 8
  Progressive disease | 5
  Inevaluable | 6
  Objective response rate (CR + PR) | 1

4. Secondary Outcome: Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of Milademetan In Participants Receiving Milademetan
Description: Plasma pharmacokinetic parameters of DS-3032a were calculated using noncompartmental methods.
Time Frame: Escalation:Cycle 1,Days 1,2,8,15,18-21 Predose,0.5,1,2,3,6-8 hours(h);Cycle 2,Day 1 Predose,1,3,6-8h,30 days after last dose; Expansion:Cycle 1,Days 1,2,8,15,18-21 Predose,0.5,1,2,3,4,6,8h;Cycle 2,Day 1 Predose,1,2,3,4,6,8h and Day 2 (each cycle, 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 33 | 2 | 5 | 9 | 15 | 5 | 3 | 3 | 3 | 20 | 3
ng/mL | 83.1 (23.8) | 198.0 | 310.0 | 551.7 (199.5) | 1525.0 (700.0) | 1301.8 (534.6) | 567.7 (341.8) | 527.7 (211.7) | 622.0 (182.8) | 757.3 (298.6) | 899.3 (466.0) | 978.0 (572.6) | 1625.4 (587.9) | 2649.7 (2160.6)

5. Secondary Outcome: Pharmacokinetic Parameter Area Under the Curve (AUC) of Milademetan In Participants Receiving Milademetan
Description: Area under the curve from time 0 to 24 hours (AUC0-24), time 0 to infinity (AUCinf), and to the last measurable concentration (AUClast). Plasma pharmacokinetic parameters of DS-3032a were calculated using noncompartmental methods.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 33 | 2 | 5 | 9 | 15 | 5 | 3 | 3 | 3 | 20 | 3
ng*h/mL
  AUC0-24: number analyzed (Participants) | 3 | 1 | 1 | 25 | 2 | 4 | 7 | 13 | 4 | 3 | 2 | 2 | 15 | 2
  AUC0-24 | 934.0 (58.9) | 2211.0 | 2930.4 | 7421.2 (3183.6) | 21386.7 (8068.1) | 17747.4 (7912.1) | 7828.7 (4229.9) | 7080.0 (2891.7) | 6943.6 (1994.2) | 9752.2 (3532.0) | 15928.8 (1235.9) | 12602.8 (8527.7) | 20006.9 (7204.6) | 39118.2 (16317.6)
  AUCinf: number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  AUCinf | 1182.2 |  | 3248.4 | 3799.4 |  |  | 12586.1 |  |  |  |  |  | 18925.3 (12784.2) | 28031.5
  AUClast | 927.1 (73.0) | 1907.2 | 2864.4 | 7375.7 (2987.9) | 20547.1 (9807.2) | 18190.2 (6652.6) | 7243.8 (4546.0) | 6798.5 (2655.4) | 7334.6 (2486.1) | 9715.2 (3532.3) | 12059.1 (6183.5) | 11928.4 (5518.5) | 19619.9 (6897.2) | 24701.2 (21198.0)

6. Secondary Outcome: Pharmacokinetic Parameter Time to Reach Maximum Plasma Concentration (Tmax) of Milademetan In Participants Receiving Milademetan
Description: Plasma pharmacokinetic parameters of DS-3032a were calculated using noncompartmental methods.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 22 | 2 | 3 | 5 | 12 | 4 | 3 | 2 | 2 | 14 | 2
hours | 13.8 [9.5 to 16.9] | 9.3 [9.3 to 9.3] | 6.7 [6.7 to 6.7] | 12.9 [5.0 to 18.1] | 14.5 [14.1 to 14.9] | 13.0 [9.4 to 16.9] | 12.8 [7.8 to 41.7] | 12.1 [8.9 to 16.3] | 13.0 [12.4 to 15.9] | 13.8 [13.4 to 14.6] | 13.4 [10.1 to 16.7] | 13.1 [10.1 to 16.0] | 11.7 [2.3 to 17.3] | 7.2 [3.8 to 10.7]

7. Secondary Outcome: Pharmacokinetic Parameter Apparent Clearance (CL/F) of Milademetan In Participants Receiving Milademetan
Description: Plasma pharmacokinetic parameters of DS-3032a were calculated using noncompartmental methods.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: L/h
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
L/h | 12.7 [12.7 to 12.7] |  | 18.5 [18.5 to 18.5] | 31.6 [31.6 to 31.6] |  |  | 7.2 [7.2 to 7.2] |  |  |  |  |  | 17.8 [9.3 to 26.3] | 12.1 [12.1 to 12.1]

8. Secondary Outcome: Pharmacokinetic Parameter Elimination Terminal Half Life Half-Life (T1/2) of Milademetan In Participants Receiving Milademetan
Description: Plasma pharmacokinetic parameters of DS-3032a were calculated using noncompartmental methods.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 22 | 2 | 3 | 5 | 12 | 4 | 3 | 2 | 2 | 14 | 2
hours | 13.4 (3.7) | 9.3 | 6.7 | 12.8 (2.9) | 14.5 (0.5) | 13.1 (3.8) | 17.6 (13.6) | 12.4 (2.3) | 13.6 (1.6) | 13.9 (0.6) | 13.4 (4.7) | 13.1 (4.2) | 10.9 (3.9) | 7.2 (4.9)

9. Secondary Outcome: Mean Fold Change From Baseline in Serum MIC-1 Levels in Participants Receiving Milademetan
Description: Mean fold change in macrophage inhibitory cytokine-1 (MIC-1) levels in serum from baseline are summarized using descriptive statistics by cohort.
Time Frame: Cycle 1, Day 15 and Cycle 1, Days 18 to 21 (each cycle is 28 days)
Population: Serum MIC-1 levels were assessed in the Biomarker Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan | Expansion Cohort: 120 mg/Day Milademetan
Number analyzed (Participants) | 3 | 1 | 1 | 13 | 1 | 4 | 9 | 15 | 4 | 3 | 3 | 3 | 18 | 3 | 18
fold change
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 1 | 1 | 13 | 1 | 4 | 7 | 15 | 4 | 3 | 3 | 3 | 18 | 3 | 18
  Cycle 1, Day 15 | 1.65 (0.5) | 2.39 | 2.05 | 6.13 (3.6) | 31.03 | 18.59 (9.5) | 5.80 (2.3) | 8.71 (5.8) | 1.21 (0.2) | 1.01 (0.2) | 1.02 (0.3) | 1.35 (0.1) | 2.85 (6.4) | 1.76 (1.6) | 4.90 (3.4)
  Cycle 1, Days 18 to 21: number analyzed (Participants) | 2 | 1 | 1 | 11 | 1 | 3 | 9 | 15 | 0 | 0 | 0 | 0 | 2 | 0 | 16
  Cycle 1, Days 18 to 21 | 1.98 (1.1) | 1.69 | 2.00 | 6.17 (3.3) | 47.40 | 15.49 (10.0) | 4.99 (1.6) | 8.32 (4.9) |  |  |  |  | 21.50 (14.6) |  | 5.48 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening until end of study, up to approximately 7 years 4 months.
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that emerged during the treatment period (from first dose date until 30 days after the last dosing date), having been absent at pretreatment; or reemerged during treatment, having been present at baseline, but stopped prior to treatment; or worsened in severity after starting treatment relative to the pretreatment state, when the AE was continuous.
Arm/Group | Cohort 1: 15 mg/Day Milademetan | Cohort 2: 30 mg/Day Milademetan | Cohort 3: 60 mg/Day Milademetan | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort | Cohort 5: 240 mg/Day Milademetan | Cohort 6: 160 mg/Day Milademetan | Cohort 7b: 90 mg/Day Milademetan | Cohort 8c: 90 mg/Day Milademetan | Cohort 9d: 120 mg/Day Milademetan | Cohort 10e: 120 mg/Day Milademetan | Cohort 11e: 200 mg/Day Milademetan | Cohort 12d: 200 mg/Day Milademetan | Cohort 13e: 260 mg/Day Milademetan | Cohort 14e: 340 mg/Day Milademetan
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/1 | 3/33 | 0/2 | 0/5 | 0/9 | 1/15 | 0/6 | 0/3 | 0/3 | 0/3 | 3/20 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/1 | 11/33 | 1/2 | 2/5 | 3/9 | 2/15 | 0/6 | 2/3 | 0/3 | 0/3 | 4/20 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/1 | 33/33 | 2/2 | 5/5 | 9/9 | 15/15 | 6/6 | 3/3 | 3/3 | 3/3 | 20/20 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 15 mg/Day Milademetan (N=3) | Cohort 2: 30 mg/Day Milademetan (N=1) | Cohort 3: 60 mg/Day Milademetan (N=1) | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort (N=33) | Cohort 5: 240 mg/Day Milademetan (N=2) | Cohort 6: 160 mg/Day Milademetan (N=5) | Cohort 7b: 90 mg/Day Milademetan (N=9) | Cohort 8c: 90 mg/Day Milademetan (N=15) | Cohort 9d: 120 mg/Day Milademetan (N=6) | Cohort 10e: 120 mg/Day Milademetan (N=3) | Cohort 11e: 200 mg/Day Milademetan (N=3) | Cohort 12d: 200 mg/Day Milademetan (N=3) | Cohort 13e: 260 mg/Day Milademetan (N=20) | Cohort 14e: 340 mg/Day Milademetan (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 15 mg/Day Milademetan (N=3) | Cohort 2: 30 mg/Day Milademetan (N=1) | Cohort 3: 60 mg/Day Milademetan (N=1) | Cohort 4: 120 mg/Day Milademetan + Expansion Cohort (N=33) | Cohort 5: 240 mg/Day Milademetan (N=2) | Cohort 6: 160 mg/Day Milademetan (N=5) | Cohort 7b: 90 mg/Day Milademetan (N=9) | Cohort 8c: 90 mg/Day Milademetan (N=15) | Cohort 9d: 120 mg/Day Milademetan (N=6) | Cohort 10e: 120 mg/Day Milademetan (N=3) | Cohort 11e: 200 mg/Day Milademetan (N=3) | Cohort 12d: 200 mg/Day Milademetan (N=3) | Cohort 13e: 260 mg/Day Milademetan (N=20) | Cohort 14e: 340 mg/Day Milademetan (N=3)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 22 | 2 | 5 | 7 | 13 | 4 | 1 | 2 | 3 | 16 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 16 | 1 | 3 | 4 | 7 | 0 | 1 | 1 | 1 | 9 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 10 | 2 | 3 | 2 | 4 | 2 | 1 | 1 | 1 | 11 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 7 | 1 | 0 | 4 | 5 | 2 | 1 | 1 | 0 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 5 | 0 | 2 | 1 | 4 | 0 | 1 | 0 | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 25 | 1 | 4 | 5 | 13 | 2 | 1 | 1 | 2 | 11 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 16 | 1 | 3 | 4 | 9 | 2 | 0 | 2 | 2 | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 | 1 | 5 | 5 | 9 | 1 | 1 | 1 | 0 | 7 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 | 1 | 4 | 4 | 6 | 1 | 0 | 0 | 0 | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 18 | 2 | 4 | 4 | 10 | 4 | 2 | 1 | 2 | 10 | 2
Oedema peripheral (General disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 1 | 3 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 10 | 2 | 5 | 5 | 7 | 1 | 1 | 0 | 0 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 5 | 1 | 1 | 2 | 5 | 3 | 0 | 0 | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 4 | 0 | 2 | 3 | 6 | 1 | 0 | 0 | 1 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 7 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 4 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 1 | 1 | 2 | 4 | 2 | 1 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tunnel vision (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver palpable subcostal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte percentage increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food aversion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimination increased (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blindness transient (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urgency hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT01877382/Prot_SAP_000.pdf